CLINICAL TRIAL: NCT01334294
Title: Home Vision Monitoring Using the ForeseeHome Device Following Treatment of Neovascular AMD
Brief Title: Home Vision Monitoring Using the ForeseeHome Device Following Treatment of Neovascular Age Related Macular Degeneration
Acronym: CNV
Status: Completed | Type: Observational
Sponsor: Notal Vision Ltd. (Industry)
Responsible Party: Sponsor
Organization: Notal Vision Inc. (Industry)
Other Study IDs: PT US 001.2
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Age Related Macular Degeneration; Choroidal Neovascularization
Keywords: CNV; AMD
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1. Received therapy for CNV
  Interventions: Device: ForeseeHome

INTERVENTIONS:
Device: ForeseeHome — The ForeseeHomeTM device, was designed to identify central and paracentral irregularities (vision abnormalities) in the visual field, most commonly associated with exudative macular degeneration.

SUMMARY:
ForeseeHome, an FDA-approved home device, was specifically designed for unsupervised Preferential-Hyperacuity-Perimeter (PHP) testing of Age Related Macular Degeneration (AMD) patients at home by characterizing central and paracentral metamorphopsia . The purpose of the current study is to evaluate if, in post-treatment patients, PHP parameters as measured with the ForeseeHome are in agreement with clinical decisions and retinal characteristics as measured with optical coherence tomography (OCT).

ELIGIBILITY:
Inclusion Criteria:

1. Received intravitreal antiangiogenic therapy for CNV in the study eye (SE), within 2-12 months prior to the study
2. Last diagnosis was, and current diagnosis is, no CNV activity in SE eye
3. Current plan in SE is clinical examination as standard care but at intervals of not more than 8 weeks.
4. Visual acuity of 20/80 or better in SE
5. Are capable and agree to sign a consent form and participate in the study
6. Age > 55 year of age
7. Are able to use a standard computer mouse correctly and without assistance
8. Have a working telephone landline at the main residence (cellular communication maybe available for the study, and then eliminate this requirement)
9. Clear view of the macular area on fundus photography
10. Are willing to give their name and contact information to Notal Vision, supplier of the device, so that the company can provide direct services if needed (e.g., assist in using the home device, report the frequency of usage, coordinate replacement of devices in case of a technical problems, etc.)
11. Agree to be examined by an ophthalmologist if SE shows symptoms of changes during the study
12. Have a US address and do not plan on traveling abroad during the study period
13. Fluent in English
14. Perform a reliable ForeseeHome test during the enrollment visit

Exclusion Criteria:

1. Evidence of macular disease other than AMD or glaucoma in SE
2. Presence of any significant media opacity that precludes a clear view of the macular area as identified in SE by biomicroscopy
3. Any non-macular related ocular surgery performed within 3 months prior to study entry in SE
4. Participant are not enrolled in another stuy that could affect the interval between clinical examinations, or the frequency of use of the ForeseeHome device

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Wet AMD
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Assess the accuracy of the ForeseeHome to detect reactivation of CNV following successful treatment with Anti-VEGF | 1 year

SECONDARY OUTCOMES:
Evaluate the correlation between PHP measures and OCT measures | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mark Michels, MD, Principal Investigator — Retina care specialists
Locations (3):
- United States (3):
  - Retina Care specisalists, Palm Beach Gardens, Florida
  - Elman retina group, Baltimore, Maryland
  - Pepose Vision Institute, St Louis, Missouri